CLINICAL TRIAL: NCT00401310
Title: A Phase IIa Randomized, Double-Blind, Parallel-Groups, Placebo Controlled Clinical Trial to Study the Efficacy and Safety of MK0724 Intravenous Infusion on the Amelioration of Neurological Damage and Recovery From Middle Cerebral Artery Ischemic Stroke
Brief Title: The Efficacy and Safety of MK0724 IV for Improvement of Neurological Damage and Recovery From Middle Cerebral Artery Ischemic Stroke (0724-018)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination date was 20-Oct-2008. Subjects were monitored during the post treatment 90 day follow-up period (per protocol) resulting in LPLV 19-Jan-2009.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0724-018; 2006_559
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Middle Cerebral Artery Stroke
MeSH Terms: conditions — Infarction, Middle Cerebral Artery

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo
- 2 (Experimental): MK0724
  Interventions: Drug: Comparator: MK0724

INTERVENTIONS:
Drug: Comparator: Placebo — Placebo IV infusions 1hr/daily over 7 days.
  Arms: 1
Drug: Comparator: MK0724 — MK0724 8 mg/kg/hr 1 hr/daily over 7 days.
  Arms: 2

SUMMARY:
The safety and efficacy of MK0724 will be assessed in patients with acute middle cerebral artery stroke using the Action Reach Arm Test (ARAT). This test allows measurement of a specific functional deficit and subsequent recovery correlating with the specific area of stroke in the brain.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 yrs of age inclusive
* Patient is able to receive IV infusion 8-36 hours after stroke onset
* Baseline NIHSS of 6-18 inclusive

Exclusion Criteria:

* Patient had another stroke within 3 months preceding current stroke, patient's stroke is of origin other than MCA (e.g., non-ischemic, hemorrhage), significant cerebral edema, abnormal liver enzymes and abnormal renal and hepatic functions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test score | At 90 days

SECONDARY OUTCOMES:
Scores on the Stroke Arm Strength question, modified Rankin, and Barthel Index. | At 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC